CLINICAL TRIAL: NCT03856398
Title: The Rigid Fiberscope With a Flexible Tip C-MAC®VS in the Real Anaesthesia World: A Clinical Observation of Intubation Success and Complications
Brief Title: C-MAC VS Clinical Observation
Status: Terminated | Type: Observational
Why Stopped: not sufficient enrolment possible
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01452
Record Dates: First submitted 2018-11-09; First posted 2019-02-27 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Intubation Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: C- MAC VS — C-MAC VS, Karl Storz AG, 78532 Tuttlingen, Germany It has a flexible tip and a distal angular offset, in which the camera and light sources are integrated. It can be aligned (up to 60°) to the patient's anatomical structures to facilitate intubation.

SUMMARY:
During orotracheal intubation failure in securing an airway can result in serious oxygenation problems.

Beside the classic laryngoscopes and fibreoptic scopes, devices with high-resolution video cameras placed in the tip of the devices, were developed and attained in daily routines. Studies and case reports reveal them to be superior in both normal and difficult intubation, especially improving the first-attempt success rate.

Latest advancements of the Bonfils fiberscope resulted in the C-MAC VS, which combines rigid and semi-rigid abilities to a rigid video stylet with a flexible tip. Because of its front positioned high-resolution camera resulting in an indirect visualization, it may also have the benefits of video laryngoscopes.

Very little data is available on larger numbers of use and the investigators do not know about rare side effects and complications with the use of the device, such as esophageal intubations. Due to its direct view and positioning on vocal cord level, the investigators expect a similar or even lower rate of endotracheal intubation, using the C-MAC VS.

The investigators therefore plan to analyze the use of the C-MAC VS regarding its efficiency and safety during airway management in everyday clinical practice. This should provide the evidence about safe use, possible risk factors, rare complications and adverse events, as well as the preferred clinical airway situations to use the C-MAC VS.

DETAILED DESCRIPTION:
Orotracheal intubation is a core competence in anesthesia and emergency medicine. Failure in securing an airway can result in hypoxemia, aspiration, neurologic damage, cardiovascular complications, and death. Difficult anatomic structures, upper airway abnormalities, or airway trauma bear the risk of failed intubation inability to ventilate the lungs that furthermore results in oxygenation failure.

Literature tells that the rate of unexpected difficult intubations ranges from 5 to 10%, mostly corresponding to a Cormack/Lehane grade (C&L) 3 or 4.

Beside the classic laryngoscopes and fibreoptic scopes, devices with high-resolution video cameras placed in the tip of the devices, were developed and attained in daily routines. Studies and case reports reveal them to be superior in both normal and difficult intubation, especially improving the first-attempt success rate.

Rigid fiber-optic scopes may reduce intubation time and their use may result in a higher success rate. A study with 216 Patients using the Bonfils fiberscope for airway management, showed a success rate up to 98,4. Looking at the complication rates, upper airway trauma in normal patients after direct laryngoscopy with a Macintosh blade has been reported up to 6.9% and can be reduced by using a video laryngoscope.

Latest advancements of the Bonfils fiberscope resulted in the C-MAC VS, which combines rigid and semi-rigid abilities to a rigid video stylet with a flexible tip. Because of its front positioned high-resolution camera resulting in an indirect visualization, it may also have the benefits of video laryngoscopes.

But data about this new tool is rare, because this device is recently licensed. Very little data is available on larger numbers of use and the investigators do not know about rare side effects and complications with the use of the device, such as esophageal intubations.

Due to its direct view and positioning on vocal cord level, the investigators expect a similar or even lower rate of endotracheal intubation using the C-MAC VS.

The investigators therefore plan to analyze the use of the C-MAC VS regarding its efficiency and safety during airway management in everyday clinical practice. This prospective observational trial should provide the evidence about safe use, possible risk factors, rare complications and adverse events, as well as the preferred clinical airway situations to use the C-MAC VS.

The investigators will check for given general research consent. All airway management procedures and the recorded data are daily clinical routine. No experimental intervention will take place, there is no change in usual clinical practice and therefore patient's safety will not be altered by participating in the study.

The study will end when the tracheal tube is placed properly and the airway is secured. On the day after surgery the investigators will visit the patient as usually after each anesthesia to obtain follow up data. In case of a complication the patient will be followed up until the problem is cured or solved.

ELIGIBILITY:
Inclusion Criteria:

* Patients for elective and emergency surgery who have at least one predictor for difficult airway management, which are: Mallampati score >2, mouth opening <4cm, thyromental distance <6cm, head & neck movements <90°, short neck, reduced reclination.
* Patients who signed general research consent in Switzerland.

Exclusion Criteria:

* Patients under the age of 18 years
* Personnel at the study site not available of not sufficient ted in the device.
* Expected impossible mask ventilation
* High risk of aspiration (requiring rapid sequence induction intubation)
* Intracranial surgery
* Limited knowledge of German language or refusing general consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing general anaesthesia for elective procedures at the Bern University Hospital will be screened using the Anesthesia Information System (AIS). Patients that meet the inclusion criteria, we will visited to confirm that and the given general consent.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
First-attempt oro-tracheal intubation success rate in percentage | The overall rate of successful intubation at first attempt. The study will end when the tracheal tube is placed properly and the airway is secured (the first attempt should not pass 120 seconds)
  Rate of a successful intubation at first attempt

SECONDARY OUTCOMES:
Overall success rate | Intraoperative (The study will end when the tracheal tube is placed properly and the airway is secured.)
  The overall rate of successful intubation.
Number of attempts | Intraoperative (Starts when the device is inserted in the patients mouth and ends when the airway is secured.)
  The total number of attempts needed for the intubation in each study session
Difficulty of intubation | Starts when the device is inserted in the patients mouth and ends when the airway is secured. Estimated time: 120 seconds
  It can range from very easy to very difficult
Preferred method used to lift the tongue ventral to increase space in the oral cavity and the approach | The beginning of the intubation procedure, when the device is inserted in the patients mouth. Estimated time 120 seconds
  The method can include using finger, laryngoscope, spatula or other. A medial, retromolar right side and retromolar left side approach can be performed.
Tube size used | Baseline
  Variations of tube sizes that will be used. It is chosen because of the patients size.
Time of the intubation procedure | Starts when the device is inserted in the patients mouth and ends when the airway is secured. Estimated time: 120 seconds
  The procedure starts as soon as the tip of the device passes patients lips and ends when a first recording of the endtidal carbon dioxide is shown.
Intubation interim times | The interim times need to be as short as possible. The estimated time for intubation: 120 seconds.
  Interim times until the device is completely out of tube
An alternative method to establish a patent airway | Starts when the device is inserted in the patients mouth and ends when the airway is secured. Estimated time for intubation: 120 seconds
  If intubation is not possible with the Intubations Device C-MAC® VS Video Stylet ,a different device has to be used for intubation. Alternative device: flexible laryngoscope,C-MAC Videolaryngoskop,Macintosh or LAMA.
Possible problems with C-MAC VS | If any problems occur during the preparations or during intubation itself which starts when the device is inserted in the patients mouth and ends when the airway is secured. Estimated time for intubation: 120 seconds
  Adverse Events, technical problems with the device
Complications during intubation | Starts when the device is inserted in the patients mouth and ends when the airway is secured. Estimated time: 120 seconds
  For example bleeding, laryngospasm, edema, swelling and other can be complications during intubation.
Airway ratings (Cormack- Lehane and POGO) | The ratings are made during the process of intubation, so when the the device is inserted in the patients mouth and ends when the airway is secured. Estimated time for intubation: 120 seconds
  Cormack- and Lehane is used to classify the laryngeal view, POGO stands for percentage of glottic opening

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, Prof., MD, Principal Investigator — Department of Anaesthesiology and Pain Therapy, Bern University Hospital
Locations (1):
- Bern University Hospital and University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mort TC. Emergency tracheal intubation: complications associated with repeated laryngoscopic attempts. Anesth Analg. 2004 Aug;99(2):607-13, table of contents. doi: 10.1213/01.ANE.0000122825.04923.15. PMID 15271750
- [Background] Peterson GN, Domino KB, Caplan RA, Posner KL, Lee LA, Cheney FW. Management of the difficult airway: a closed claims analysis. Anesthesiology. 2005 Jul;103(1):33-9. doi: 10.1097/00000542-200507000-00009. PMID 15983454
- [Background] Williams KN, Carli F, Cormack RS. Unexpected, difficult laryngoscopy: a prospective survey in routine general surgery. Br J Anaesth. 1991 Jan;66(1):38-44. doi: 10.1093/bja/66.1.38. PMID 1997057
- [Background] Maassen R, Lee R, van Zundert A, Cooper R. The videolaryngoscope is less traumatic than the classic laryngoscope for a difficult airway in an obese patient. J Anesth. 2009;23(3):445-8. doi: 10.1007/s00540-009-0780-1. Epub 2009 Aug 14. PMID 19685133
- [Background] Choi JW, Kim JA, Jung HJ, Kim WH. Tracheal Intubation with a McGrath(R) Series 5 Video Laryngoscope by Novice Personnel in a Cervical-immobilized Manikin. J Emerg Med. 2016 Jan;50(1):61-6. doi: 10.1016/j.jemermed.2015.06.079. Epub 2015 Oct 1. PMID 26432080
- [Background] Burdett E, Ross-Anderson DJ, Makepeace J, Bassett PA, Clarke SG, Mitchell V. Randomized controlled trial of the A.P. Advance, McGrath, and Macintosh laryngoscopes in normal and difficult intubation scenarios: a manikin study. Br J Anaesth. 2011 Dec;107(6):983-8. doi: 10.1093/bja/aer295. Epub 2011 Sep 22. PMID 21940397
- [Background] Kory P, Guevarra K, Mathew JP, Hegde A, Mayo PH. The impact of video laryngoscopy use during urgent endotracheal intubation in the critically ill. Anesth Analg. 2013 Jul;117(1):144-9. doi: 10.1213/ANE.0b013e3182917f2a. Epub 2013 May 17. PMID 23687228